CLINICAL TRIAL: NCT04041219
Title: Use of Sublingual Tacrolimus in Adult Blood and Marrow Transplant Patients: a Pilot Study
Brief Title: Use of Sublingual Tacrolimus in Adult Blood and Marrow Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Heather P May, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000181
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Immunosuppression; Stem Cell Transplant; Bone Marrow Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic blood or marrow transplantation (Experimental): Subjects undergoing allogeneic blood or marrow transplantation (BMT) at Mayo Clinic in Rochester Minnesota
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Recommended starting dose will be in accordance with the established protocol (0.04 mg/kg/dose of ideal body weight), initially administered sublingually for four consecutive doses.
Drug: Tacrolimus — Recommended starting dose will be in accordance with the established protocol (0.04 mg/kg/dose of ideal body weight), oral administration after sublingual four consecutive doses

SUMMARY:
Researchers are trying to learn more about using sublingual (absorption under the tongue) tacrolimus in blood and marrow transplant patients.

DETAILED DESCRIPTION:
Initial doses will be given via sublingual route and a steady state trough level will be collected after 4 consecutive doses. Participants will then switched to oral tacrolimus, the dose adjusted for a goal trough 8-12ng/mL, and another steady state trough will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be identified from within the adult allogeneic BMT program at Mayo Clinic in Rochester, Minnesota
* Adults prescribed tacrolimus for treatment or prevention of Graft Versus Host Disease (GVHD)

Exclusion Criteria:

* Vulnerable populations
* Patients with contraindications to tacrolimus, inclusive of hypersensitivity, history of posterior reversible encephalopathy syndrome or calcineurin-inhibitor induced thrombotic microangiopathy
* Lacking the capacity to consent in English and declining to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather May, Pharm. D., R. Ph., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] May HP, Bartoo GT, Wolf RC, Shah MV, Litzow MR, Hogan WJ, Alkhateeb H. Use of sublingual tacrolimus in adults undergoing hematopoietic cell transplant: A pilot study. J Oncol Pharm Pract. 2022 Mar;28(2):387-394. doi: 10.1177/1078155221995230. Epub 2021 Feb 16. PMID 33593135
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic Blood or Marrow Transplantation: Subjects who had allogeneic blood or marrow transplantation (BMT) at Mayo Clinic in Rochester Minnesota
  Tacrolimus: Recommended starting dose was in accordance with the established protocol (0.04 mg/kg/dose of ideal body weight), initially administered sublingually for four consecutive doses.
  Tacrolimus: Recommended starting dose was in accordance with the established protocol (0.04 mg/kg/dose of ideal body weight), oral administration after sublingual four consecutive doses
Period: Overall Study
Arm/Group | Allogeneic Blood or Marrow Transplantation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Blood or Marrow Transplantation
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [51 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Hematologic Diagnosis of Acute myeloid leukemia [Count of Participants; unit: Participants] | 6
Hematologic Diagnosis of Myelodysplastic syndrome [Count of Participants; unit: Participants] | 2
Hematologic Diagnosis of Other [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Tacrolimus Sublingual Trough Level
Description: Trough level is the lowest concentration in the patient's bloodstream and was collected after four consecutive sublingual doses. Measured as ng/mL.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Allogeneic Blood or Marrow Transplantation
Number analyzed (Participants) | 10
ng/mL | 11.3 [6 to 17.4]

2. Secondary Outcome: Median Sublingual (SL) to Oral (PO) Ratio
Description: Total daily dose will be divided by the corresponding trough whole blood concentration for each route of administration to determine the dosing ratio of SL:PO. [(daily doseSL/blood concentrationSL)/(daily dosePO/blood concentrationPO)] for each individual participant.
Time Frame: 14 days
Measure: Median (Full Range); unit: ratio
Arm/Group | Allogeneic Blood or Marrow Transplantation
Number analyzed (Participants) | 10
ratio | 1.02 [0.57 to 1.92]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from three days prior to transplant to end study for a total of approximately 30 days for each subject.
Arm/Group | Allogeneic Blood or Marrow Transplantation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT04041219/Prot_SAP_000.pdf